CLINICAL TRIAL: NCT03616652
Title: Non-deceptive Application of Placebos in Insomnia
Acronym: NAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-43k
Record Dates: First submitted 2018-07-20; First posted 2018-08-06 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-deceptive placebo group (additional information) (Experimental): Participants receive a placebo pill and are told that it is placebo. They receive additional information about the power of placebo effects via a film sequence before they take the placebo.
  Interventions: Drug: Placebo; Other: Film sequence
- Non-deceptive placebo group (no additional information) (Placebo Comparator): Participants receive a placebo pill and are told that it is placebo. They do not receive additional information about placebo effects. Instead, they watch a neutral film sequence about sleep.
  Interventions: Drug: Placebo; Other: Film sequence

INTERVENTIONS:
Drug: Placebo — Placebo pill
Other: Film sequence — The experimental group watches a film about the power of placebo effects.
  Arms: Non-deceptive placebo group (additional information)
Other: Film sequence — The control group watches a film about sleep.
  Arms: Non-deceptive placebo group (no additional information)

SUMMARY:
The purpose of this study is to evaluate whether non-deceptive application of a placebo has an impact on subjective or objective sleep parameters in patients with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 years to 69 years
* fluent in German language
* provide written informed consent
* ability to understand the explanations and instructions given by the study physician and the investigator

Exclusion Criteria:

* evidence for sleep disorders caused by medical factors (e.g. sleep apnea, restless legs syndrome, narcolepsy, substance-induced insomnia)
* allergies to ingredients of placebo
* patients scoring below 8 or above 21 on the Insomnia Severity Index
* patients suffering from a mental disorder as verified by the SCID
* patients suffering from an acute physical illness
* nicotine consumption > 10 cigarettes/day
* unwillingness to refrain from alcohol consumption throughout the study
* change in concomitant medication regime during the last 2 weeks prior to visit 1 or after randomization
* intake of psychotropic drugs during the last 3 months prior to visit 1
* currently pregnant (verified by urine pregnancy test) or lactating

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Self-reported Total Sleep Time | change from baseline to 1 night after placebo intake
  assessed by sleep diary

SECONDARY OUTCOMES:
Objective Sleep Efficiency | change from baseline to 1 night after placebo intake
  assessed by actigraphy
Objective Total Sleep Time | change from baseline to 1 night after placebo intake
  assessed by actigraphy
Objective Total Sleep Time | change from baseline to 1 night after placebo intake
  assessed by polysomnography
Objective Sleep Onset Latency | change from baseline to 1 night after placebo intake
  assessed by polysomnography
Self-reported Sleep Onset Latency | change from baseline to 1 night after placebo intake
  assessed by sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Clinical Psychology and Psychotherapy, Department of Psychology, Philipps University Marburg
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany